CLINICAL TRIAL: NCT04693247
Title: An Exploratory Study in Healthy Adult Volunteers to Evaluate the Best Corrected Visual Acuity (BCVA) Performance of a Handheld Device Compared With a Standard Eye Care Diagnostic Device in Measuring Ophthalmic Refraction
Brief Title: Handheld Device Compared With a Standard Eye Care Diagnostic Device in Measuring Ophthalmic Refraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: EyeQue Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: EYEQUE - 004
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Refractive Errors; Vision Disorders
MeSH Terms: conditions — Refractive Errors; Vision Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Tester and subject for BCVA are masked as to which device and trial frames are from.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Refraction with a Hand-held Refraction Device (Active Comparator): This is the device that will be compared to a standard device.
  Interventions: Device: EQ103
- Autorefractor (Other): Standard Device
  Interventions: Device: EQ103

INTERVENTIONS:
Device: EQ103 — Refraction device

SUMMARY:
This study is exploratory and examines whether the best-corrected visual acuities (BCVA's) from trial frames created with the refraction results obtained from a novel handheld optical device yields results similar to the ophthalmic refraction obtained from an autorefractor in healthy volunteers age stratum of 18 through 65 years.

DETAILED DESCRIPTION:
This study is exploratory and examines whether the best-corrected visual acuities (BCVA's) from trial frames created with the refraction results obtained from a novel handheld optical device yields results similar to the ophthalmic refraction obtained from an autorefractor in healthy volunteers age stratum of 18 through 65 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Ages =>18 y.o. and =<65 y.o.
* Binocular vision
* Willing and able to give informed consent and follow all study procedures and requirements
* Fluent in English

Exclusion Criteria:

* Has been diagnosed within 4 weeks, or currently has signs or symptoms, of COVID-19.
* Has traveled outside the country within the last 4 weeks.
* At the discretion of the investigator: Age strata has achieved minimum evaluable population.
* Spherical correction > +8 or < -10
* Using anticholinergic medications (including first-generation antihistamines) or other medications known to affect visual acuity within the greater of 3 days or 5 half-lives prior to enrolling in this study
* Using an investigational drug or approved therapy for investigational use within the greater of 3 days or 5 half-lives prior to enrolling in this study
* Has initiated any new medication in the past 2 weeks that, in the best medical judgment of the investigator, would impact their participation in the study or ability to use the EyeQue EQ103 device
* Any self-reported mental illness or condition, including but not limited to:

claustrophobia, fear of simulators, nyctophobia.

* Any self-reported neurological diseases, including but not limited to: epilepsy, Alzheimer's, nystagmus

Per subject self-reporting: eye disease, including but not limited to:

* Glaucoma
* Cataracts
* Macular degeneration
* Eye infection (by self-report or observation)
* Keratoconus
* Diabetic neuropathy/retinopathy
* Cytomegalovirus retinitis
* Color blindness (any color deficiency)
* Diabetic macular edema
* Amblyopia
* Chronic or acute uveitis
* Strabismus
* Astigmatism > 3 diopters
* Macular hole

Subjects that:

* Lack physical dexterity to properly operate the EyeQue device.
* Lack the ability to follow instruction
* Lack a command of the English language
* Lack binocular vision
* Are colorblind
* Had eye surgery within the last 12 months (including Lasik)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2023-06-21 (Estimated); Study Completion 2023-06-21 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity (BCVA) for both eyes EQ103 vs Autorefractor for all participants | Day 1
  Tendency of, or achieving, statistical non-inferiority of EyeQue EQ103 BCVA's (reading an EDTRS chart) for each eye from (pooled) trial frames created with the refraction values compared with those of an autorefractor analyzed with all age groups.

SECONDARY OUTCOMES:
Best corrected visual acuity (BCVA) for both eyes EQ103 vs Autorefractor examining age groupings | Day 1
  Tendency of, or achieving, statistical non-inferiority of EyeQue EQ103 BCVA's (reading an EDTRS chart for each eye (pooled) from trial frames created with the refraction values compared with those of an autorefractor analyzed within the following age strata.
  o Age Groups: 18 - 29, 30 - 44, 45 - 65
Best corrected visual acuity (BCVA) for worse eye: EQ103 vs Autorefractor for all subjects and age groupings | Day 1
  Tendency of, or achieving, statistical non-inferiority of EyeQue EQ103 BCVA's (reading an EDTRS chart for worse eye from trial frames created with the refraction values compared with those of an autorefractor analyzed within the following age strata.
  o Age Groups: All, 18 - 29, 30 - 44, 45 - 65

CONTACTS AND LOCATIONS:
Locations (1):
- EyeQue, Newark, California, United States